CLINICAL TRIAL: NCT02025621
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Levosimendan in Patients With Left Ventricular Systolic Dysfunction Undergoing Cardiac Surgery Requiring Cardiopulmonary Bypass
Brief Title: Levosimendan in Patients With Left Ventricular Systolic Dysfunction Undergoing Cardiac Surgery On Cardiopulmonary Bypass
Acronym: LEVO-CTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNX-LVO-01
Record Dates: First submitted 2013-12-18; First posted 2014-01-01 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Bypass Grafting; Mitral Valve Surgery; Low Cardiac Output Syndrome
Keywords: coronary artery bypass grafting; CABG; mitral valve; LCOS; low cardiac output syndrome; levosimendan
MeSH Terms: conditions — Cardiac Output, Low | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Experimental): levosimendan 0.2 µg/kg/min for first hour, followed by 0.1 µg/kg/min for an additional 23 hours
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): placebo 0.2 µg/kg/min for first hour, followed by 0.1 µg/kg/min for an additional 23 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan
  Other Names: Simdax
  Arms: Levosimendan
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
A study to evaluate levosimendan compared with placebo in reducing the composite event rate of all-cause death, perioperative MI, need for new dialysis, or use of mechanical assist (IABP, LVAD or ECMO) in subjects with reduced ejection fraction undergoing cardiac surgery on cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
This study is being done to evaluate the efficacy of levosimendan compared with placebo in reducing the co-primary endpoints of 30-day composite of all-cause death or use of mechanical assist device (IABP, LVAD or ECMO) or the composite event rate of all-cause death, perioperative MI, need for dialysis, or use of mechanical assist (IABP, LVAD or ECMO) in subjects with reduced ejection fraction undergoing cardiac surgery on CPB.

ELIGIBILITY:
Inclusion Criteria:

* Documented LVEF ≤35% measured by ventriculogram, echocardiogram (ECHO), nuclear scan, or MRI within 60 days before surgery.
* Scheduled or urgent 1) CABG surgery, 2)CABG with aortic valve surgery, 3) CABG with mitral valve surgery, or 4) mitral valve surgery with or without other valves
* Surgery will employ CPB pump
* Signed (by the subjects or their legally acceptable representatives) informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Restrictive or obstructive cardiomyopathy, constrictive pericarditis, restrictive pericarditis, pericardial tamponade, or other conditions in which cardiac output is dependent on venous return.
* Evidence of systemic bacterial, systemic fungal, or viral infection within 72 hours before surgery.
* Dialysis at randomization (either hemodialysis, peritoneal dialysis, continuous venovenous hemofiltration, or ultrafiltration).
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2.
* Weight ≥ 170 kg.
* Patients whose SBP cannot be managed to ensure SBP > 90 mmHg at initiation of study drug.
* Heart rate ≥ 120 bpm, persistent for at least 10 minutes screening and unresponsive to treatment.
* Hemoglobin < 80 g/L.
* Serum potassium < 3.5 mmol/L and > 5.5 mmol/L at baseline.
* A history of Torsades de Pointes.
* Mechanical assist device (IABP, LVAD, ECMO) in the patient at the start of surgery or pre-planned to be inserted during surgery before coming off CPB.
* Patients with aortal femoral occlusive disease that would prohibit use of IABP unless VAD or ECMO not available.
* Liver dysfunction Child Pugh Class B or C
* Patients having severely compromised immune function
* Pregnant, suspected to be pregnant, or breast-feeding.
* Received an experimental drug or used an experimental medical device in previous 30 days.
* Known allergic reaction or sensitivity to Levosimendan or excipients.
* Received commercial Levosimendan within 30 days before the planned start of study drug.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra Mehta, MD, Principal Investigator — Duke Clinical Research Institute; John Alexander, MD, Study Chair — Duke Clinical Research Institute
Locations (60):
- United States (49):
  - University of Alabama at Burlington Hospital, Burlington, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Mercy General Hospital, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Redmond Regional Medical Center, Rome, Georgia
  - Northwestern University Hospital, Evanston, Illinois
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Iowa Heart Center/ Mercy Medical Center, West Des Moines, Iowa
  - University of Louisville Hospital, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - St. Joseph's Mercy Hospital, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - St. Peter's Hospital, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Saint Francis Hospital/The Heart Center, Roslyn, New York
  - Mission Hospital, Asheville, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Duke University Hospital, Raleigh, North Carolina
  - The Christ's Hospital; Lindner Clinical Trial Center, Cincinnati, Ohio
  - Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Thomas Heart, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Hospital, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Franciscan Health System Res. Center, Tacoma, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Jubilee Hospital (Vancouver Island Health Authority), Victoria, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface Hospital, Winnepeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Center, University Hospital, London, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre-Royal Victoria Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institute universitaire de cardiologie et pneumologie de Quebec, Québec

REFERENCES:
- [Derived] Verma S, Rathwell S, Fremes S, Zheng Y, Mehta R, Lopes RD, Alexander JH, Goodman SG, Diepen SV; LEVO-CTS investigators. Associated factors and clinical outcomes in mechanical circulatory support use in patients undergoing high risk on-pump cardiac surgery: Insights from the LEVO-CTS trial. Am Heart J. 2022 Jun;248:35-41. doi: 10.1016/j.ahj.2022.02.013. Epub 2022 Mar 7. PMID 35263653
- [Derived] Mehta RH, Leimberger JD, van Diepen S, Meza J, Wang A, Jankowich R, Harrison RW, Hay D, Fremes S, Duncan A, Soltesz EG, Luber J, Park S, Argenziano M, Murphy E, Marcel R, Kalavrouziotis D, Nagpal D, Bozinovski J, Toller W, Heringlake M, Goodman SG, Levy JH, Harrington RA, Anstrom KJ, Alexander JH; LEVO-CTS Investigators. Levosimendan in Patients with Left Ventricular Dysfunction Undergoing Cardiac Surgery. N Engl J Med. 2017 May 25;376(21):2032-2042. doi: 10.1056/NEJMoa1616218. Epub 2017 Mar 19. PMID 28316276
- [Derived] Mehta RH, Van Diepen S, Meza J, Bokesch P, Leimberger JD, Tourt-Uhlig S, Swartz M, Parrotta J, Jankowich R, Hay D, Harrison RW, Fremes S, Goodman SG, Luber J, Toller W, Heringlake M, Anstrom KJ, Levy JH, Harrington RA, Alexander JH; LEVO-CTS Investigators. Levosimendan in patients with left ventricular systolic dysfunction undergoing cardiac surgery on cardiopulmonary bypass: Rationale and study design of the Levosimendan in Patients with Left Ventricular Systolic Dysfunction Undergoing Cardiac Surgery Requiring Cardiopulmonary Bypass (LEVO-CTS) trial. Am Heart J. 2016 Dec;182:62-71. doi: 10.1016/j.ahj.2016.09.001. Epub 2016 Sep 9. PMID 27914501
- [Derived] Lim JY, Deo SV, Rababa'h A, Altarabsheh SE, Cho YH, Hang D, McGraw M, Avery EG, Markowitz AH, Park SJ. Levosimendan Reduces Mortality in Adults with Left Ventricular Dysfunction Undergoing Cardiac Surgery: A Systematic Review and Meta-analysis. J Card Surg. 2015 Jul;30(7):547-54. doi: 10.1111/jocs.12562. Epub 2015 May 19. PMID 25989324
- [Derived] Toller W, Heringlake M, Guarracino F, Algotsson L, Alvarez J, Argyriadou H, Ben-Gal T, Cerny V, Cholley B, Eremenko A, Guerrero-Orriach JL, Jarvela K, Karanovic N, Kivikko M, Lahtinen P, Lomivorotov V, Mehta RH, Music S, Pollesello P, Rex S, Riha H, Rudiger A, Salmenpera M, Szudi L, Tritapepe L, Wyncoll D, Owall A. Preoperative and perioperative use of levosimendan in cardiac surgery: European expert opinion. Int J Cardiol. 2015 Apr 1;184:323-336. doi: 10.1016/j.ijcard.2015.02.022. Epub 2015 Feb 24. PMID 25734940

RESULTS

PARTICIPANT FLOW:
Groups:
- Levosimendan: levosimendan 0.2 µg/kg/min for first hour, followed by 0.1 µg/kg/min for an additional 23 hours
  Levosimendan
Period: Overall Study
Arm/Group | Levosimendan | Placebo
Started | 442 | 440
Completed | 428 | 421
Not Completed | 14 | 19
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Not completed — No longer eligible | 10 | 15
Not completed — Surgery initiated before infusion | 3 | 3

BASELINE CHARACTERISTICS:
Population: Patients that received any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Levosimendan | Placebo | Total
Number analyzed (Participants) | 428 | 421 | 849
Age, Continuous [Median (Full Range); unit: years] | 65 [59 to 73] | 65 [58 to 72] | 65 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 89 | 170
  Male | 347 | 332 | 679
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 385 | 375 | 760
  Black | 21 | 23 | 44
  Asian | 9 | 10 | 19
  American Indian or Alaska Native | 2 | 4 | 6
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 5 | 7 | 12
  Not given | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 71 | 88 | 159
  United States | 357 | 333 | 690

OUTCOME MEASURES:

1. Primary Outcome: Number of Dual Efficacy Endpoint Events
Description: The all-cause death at 30 days or use of mechanical assist device (IABP, LVAD or ECMO) following the start of surgery for poor cardiac function despite inotropic support and adequate fluid replacement) through Day 5
Time Frame: 30 days
Population: mITT; population receiving any study drug
Measure: Number; unit: events
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
events | 56 | 48

2. Primary Outcome: Number of Quad Efficacy Endpoint Events
Description: Composite of all-cause death (at 30 days), or perioperative nonfatal MI [CK-MB >10xULN or >100 ng/mL, CK-MB >5xULN or 50 ng/mL with new Q wave (>0.04 seconds wide in two contiguous leads) or new left bundle branch block)] (through Day 5), or need for renal dialysis (through Day 30), or use of mechanical assist device (IABP, LVAD or ECMO) following the start of surgery for poor cardiac function despite inotropic support and adequate fluid replacement) (through Day 5)
Time Frame: 30 days
Population: mITT; population receiving any study drug
Measure: Number; unit: events
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
events | 105 | 103

3. Secondary Outcome: Duration of Intensive Care Unit/Critical or Coronary Care Unit (ICU/CCU) (Days)
Description: Duration of intensive care unit/critical or coronary care unit (ICU/CCU) length of stay (LOS) in days
Time Frame: participants will be followed for during the participant's hospital stay up to 30 days
Population: mITT; patients that received any study drug
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
days | 2.8 [1.6 to 4.8] | 2.9 [1.8 to 4.9]

4. Secondary Outcome: Incidence of Low Cardiac Output Syndrome (LCOS)
Description: Use of a mechanical cardiac assist device within 5 days after surgery, two consecutive measurements of low cardiac output (defined as a cardiac output of ≤2.0 liters per minute per square meter of bodysurface area), one measurement of low cardiac output plus the use of two or more inotropes at or beyond 24 hours after surgery, or the use of two or more inotropes at or beyond 24 hours after surgery with the indicated reason being low cardiac output.
Time Frame: 5 days
Population: mITT; patients receiving any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
Participants | 78 | 108

5. Secondary Outcome: Postoperative Use of Secondary Inotrope
Description: Use of (dobutamine, milrinone, epinephrine, dopamine) associated with index surgical procedure at 24 hours after initiation of surgery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
Participants | 235 | 264

6. Other Pre Specified Outcome: Occurrence of All-cause Mortality From Randomization Through Day 90
Time Frame: 90 days
Population: all patients receiving study drug, according to the drug actually received
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
Participants | 20 | 30

7. Other Pre Specified Outcome: Rehospitalization for Any Cause Through Day 30
Time Frame: 30 days
Population: patients receiving study drug, by study drug received
Measure: Count of Participants; unit: Participants
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 428 | 421
Participants | 54 | 48

ADVERSE EVENTS:
Time Frame: through Day 30
Arm/Group | Levosimendan | Placebo
All-Cause Mortality (participants affected / at risk) | 20/428 | 30/421
Serious Adverse Events (participants affected / at risk) | 34/428 | 37/421
Other Adverse Events (participants affected / at risk) | 238/428 | 232/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=428) | Placebo (N=421)
Cardiogenic Shock (Cardiac disorders) | 5 (5) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 6 (6)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory accidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsi (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=428) | Placebo (N=421)
Thrombocytopenia (Blood and lymphatic system disorders) | 38 (38) | 38 (38)
Anaemia (Cardiac disorders) | 35 (35) | 24 (24)
Leukocytosis (Blood and lymphatic system disorders) | 16 (16) | 23 (23)
Coagulopathy (Blood and lymphatic system disorders) | 22 (22) | 9 (9)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 12 (12) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 30 (31)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 19 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9)
Acute kidney injury (Renal and urinary disorders) | 49 (50) | 51 (54)
Urinary retention (Renal and urinary disorders) | 7 (7) | 13 (13)
Cardiogenic shock (Cardiac disorders) | 17 (17) | 15 (15)
Sinus tachycardia (Cardiac disorders) | 9 (9) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (16) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (15) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (11) | 6 (6)
Fluid overload (Metabolism and nutrition disorders) | 9 (9) | 7 (7)
Delirium (Psychiatric disorders) | 19 (21) | 12 (13)
Hypotension (Cardiac disorders) | 155 (155) | 138 (138)
Atrial fibrillation/flutter (Cardiac disorders) | 159 (159) | 134 (134)
Ventricular tachycardia/fibrillation (Cardiac disorders) | 46 (46) | 41 (41)
Stroke (General disorders) | 15 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No